CLINICAL TRIAL: NCT00882206
Title: A Therapeutic Trial of Decitabine and Vorinostat in Combination With Chemotherapy (Vincristine, Prednisone, Doxorubicin and PEG-Asparaginase) for Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LL)
Brief Title: Pre-reinductive Decitabine and Vorinostat in Relapsed Lymphoblastic Lymphoma or Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS112; 0810M50401 (Other: IRB, University of Minnesota); MT2008-29R (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; Decitabine; Doxorubicin; Imatinib Mesylate; Methotrexate; pegaspargase; Prednisone; Vincristine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine / Vorinostat (Experimental): This is a therapeutic trial investigating the combination of decitabine 15 mg/m2 and vorinostat 230 mg/m2 (maximum daily dose not to exceed 400 mg) in relapsed/refractory ALL/LL patients prior to induction chemotherapy.
  Interventions: Drug: cytarabine; Drug: decitabine; Drug: doxorubicin hydrochloride; Drug: imatinib mesylate; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: vincristine sulfate; Drug: vorinostat

INTERVENTIONS:
Drug: cytarabine — At baseline when peripheral blood draw and bone marrow aspirate performed.
  *Intrathecal Cytarabine administered dependent upon age - ranging from 30 mg to 70 mg.
  Other Names: cytosine arabinoside
Drug: decitabine — Days 1-4, 15 mg/m^2 intravenously (IV) over 1 hour
  Other Names: Dacogen(R)
Drug: doxorubicin hydrochloride — Day 5, 60 mg/m^2 intravenously (IV) over 15 minutes
  Other Names: Doxorubicin
Drug: imatinib mesylate — 340 mg/m2 by mouth every day (rounded to the nearest 100 mg) for age <18 years and 400 mg orally every day for >18 years on Days 5-33.
  Other Names: Gleevec(R)
Drug: methotrexate — **Intrathecal Methotrexate administered dependent upon age - ranging from 8 mg to 15 mg.
  Other Names: MTX
Drug: pegaspargase — 2,500 IU/m2 IM or IV q week (days 6, 12, 19, 26)
  Other Names: PEG asparaginase
Drug: prednisone — 40mg/m2/day divided BID (days 5 - 33)
Drug: vincristine sulfate — 1.5mg/m2 (max 2 mg) iv push q week (days 5, 12, 19, 26)
  Other Names: Oncovin(R)
Drug: vorinostat — Days 1-4, (230 mg/m2)orally divided twice a day (max dose 400 mg daily)
  Other Names: suberoylanilide hydroxamic acid (SAHA)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Decitabine and vorinostat may alter the cancer cells by reversing the cancer pathways needed for cell growth. Giving more than one drug (combination chemotherapy) together with decitabine and vorinostat may kill more cancer cells than with chemotherapy alone.

PURPOSE: This phase II trial is studying how well giving decitabine and vorinostat together with combination chemotherapy works in treating patients with acute lymphoblastic leukemia or lymphoblastic lymphoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Patients undergo blood and bone marrow sample collection at baseline, on day 5, Day 19 and at the end of study treatment for correlative laboratory studies. Samples are analyzed for hypermethylation at diagnosis and demethylation post-exposure with decitabine and vorinostat using LINE methylation.

OUTLINE:

Patients receive decitabine IV over 1 hour and oral vorinostat twice daily on days 1-4; vincristine sulfate IV on days 5, 12, 19, and 26; oral prednisone twice daily on days 5-33; doxorubicin hydrochloride IV over 15 minutes and cytarabine intrathecally (IT) on day 5; pegaspargase IV or intramuscularly on days 6, 12, 19, and 26; and methotrexate* IT on days 12 and 33. Patients with Philadelphia chromosome-positive disease may also receive oral imatinib mesylate once daily on days 5-33.

NOTE: *Patients with central nervous system (CNS)-positive disease also receive methotrexate IT on days 19 and 26.

Patients undergo blood and bone marrow sample collection at baseline, on day 5, Day 19 and at the end of study treatment for correlative laboratory studies.

After completion of study treatment, patients are followed for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoblastic lymphoma or acute lymphoblastic leukemia with ≥ 5% blasts in the bone marrow (M2/M3) (with or without extramedullary disease) that meets 1 of the following criteria:

  * Refractory disease/induction failure (failure to achieve initial remission after 2 lines of induction therapy)
  * Relapsed disease (in first relapse or higher)
* Central nervous system (CNS)-positive disease allowed
* Karnofsky performance status (PS) 50-100% (for patients ≥ 16 years of age) OR Lansky PS 50-100% (for patients < 16 years of age)
* Life expectancy ≥ 8 weeks
* Creatinine clearance ≥ 70 mL/min OR maximum serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (for patients 1 to 5 months of age)
  * 0.5 mg/dL (for patients 6 to 11 months of age)
  * 0.6 mg/dL (for patients 1 year of age)
  * 0.8 mg/dL (for patients 2 to 5 years of age)
  * 1.0 mg/dL (for patients 6 to 9 years of age)
  * 1.2 mg/dL (for patients 10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients ≥ 16 years of age)
* ALT < 5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN for age
* LVEF ≥ 40% by ECHO/MUGA scan
* Shortening fraction > 29% by ECHO/MUGA scan
* Able to swallow capsules
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after completion of study treatment
* No untreated positive blood cultures or progressive infections as assessed by radiographic studies
* No known allergy to any of the agents or their ingredients used in this study

  * Patients with clinically significant prior allergies to pegaspargase may be treated with asparaginase-Erwinia, if available
* Patients who cannot receive asparaginase on this study (e.g., due to prior pancreatitis, stroke, or other toxicity) are eligible provided they meet all other inclusion/exclusion criteria
* Recovered from prior therapy (defined as CTCAE v3.0 toxicity ≤ grade 1)
* More than 3 weeks since prior chemotherapy for cancer other than hydroxyurea for patients with WBC > 10,000/mm³
* At least 7 days since prior hematopoietic growth factors (14 days for pegfilgrastim)
* At least 1 month since prior biologic therapy, such as monoclonal antibodies
* At least 3 months since prior hematopoietic stem cell transplantation

Exclusion Criteria:

* Evidence of graft-versus-host disease
* Concurrent valproic acid
* Concurrent coumadin/warfarin other than a short course administered in a prophylactic setting

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Burke, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Burke MJ, Lamba JK, Pounds S, Cao X, Ghodke-Puranik Y, Lindgren BR, Weigel BJ, Verneris MR, Miller JS. A therapeutic trial of decitabine and vorinostat in combination with chemotherapy for relapsed/refractory acute lymphoblastic leukemia. Am J Hematol. 2014 Sep;89(9):889-95. doi: 10.1002/ajh.23778. Epub 2014 Jun 27. PMID 24891274

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine / Vorinostat: This is a therapeutic trial investigating the combination of decitabine 15 mg/m2 and vorinostat 230 mg/m2 (maximum daily dose not to exceed 400 mg) in relapsed/refractory ALL/LL patients prior to induction chemotherapy.
  cytarabine: At baseline when peripheral blood draw and bone marrow aspirate performed.
  *Intrathecal Cytarabine administered dependent upon age - ranging from 30 mg to 70 mg.
  decitabine: Days 1-4, 15 mg/m^2 intravenously (IV) over 1 hour
  doxorubicin hydrochloride: Day 5, 60 mg/m^2 intravenously (IV) over 15 minutes
  imatinib mesylate: 340 mg/m2 by mouth every day (rounded to the nearest 100 mg) for age <18 years and 400 mg orally every day for >18 years on Days 5-33.
  methotrexate: **Intrathecal Methotrexate administered dependent upon age - ranging from 8 mg to 15 mg.
  pegaspargase: 2,500 IU/m2 IM or IV q week (days 6, 12, 19, 26)
  prednisone: 40mg/m2/day divided BID (days 5 - 33)
  vincristine sulfate: 1.5mg/m2 (max 2 mg) iv push q week (days 5, 12,
Period: Overall Study
Arm/Group | Decitabine / Vorinostat
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine / Vorinostat
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 16 [3 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment
Description: Response includes both complete remission (defined as <5% leukemic blasts in the bone marrow) and partial remission (defined as a greater than 35% reduction in the bone marrow leukemia blast percentage at day 33)
Time Frame: Day 33
Population: The following participants were removed from the analysis: two patients had an early death; one patient had early disease progression; one patient was found to have nervous system involvement on day 5 of therapy; and one patient stopped study therapy due to toxicities.
Measure: Number; unit: participants
Arm/Group | Decitabine / Vorinostat
Number analyzed (Participants) | 8
participants | 6

2. Secondary Outcome: Level of Methylation
Description: the percentage of methylated DNA
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: percentage of DNA
Arm/Group | Decitabine / Vorinostat
Number analyzed (Participants) | 8
percentage of DNA | 84.98 (1.48)

3. Secondary Outcome: Level of Methylation
Description: the percentage of methylated DNA
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of DNA
Arm/Group | Decitabine / Vorinostat
Number analyzed (Participants) | 8
percentage of DNA | 79.82 (3.04)

4. Secondary Outcome: Level of Methylation
Description: the percentage of methylated DNA
Time Frame: Day 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of DNA
Arm/Group | Decitabine / Vorinostat
Number analyzed (Participants) | 8
percentage of DNA | 86.1 (1.87)

ADVERSE EVENTS:
Groups:
- Decitabine / Vorinostat: This is a therapeutic trial investigating the combination of decitabine 15 mg/m2 and vorinostat 230 mg/m2 (maximum daily dose not to exceed 400 mg) in relapsed/refractory ALL/LL patients prior to induction chemotherapy.
  cytarabine: At baseline when peripheral blood draw and bone marrow aspirate performed.
  *Intrathecal Cytarabine administered dependent upon age - ranging from 30 mg to 70 mg.
  decitabine: Days 1-4, 15 mg/m^2 intravenously (IV) over 1 hour
  doxorubicin hydrochloride: Day 5, 60 mg/m^2 intravenously (IV) over 15 minutes
  imatinib mesylate: 340 mg/m2 by mouth every day (rounded to the nearest 100 mg) for age <18 years and 400 mg orally every day for >18 years on Days 5-33.
  methotrexate: **Intrathecal Methotrexate administered dependent upon age - ranging from 8 mg to 15 mg.
  pegaspargase: 2,500 IU/m2 IM or IV q week (days 6, 12, 19, 26)
  prednisone: 40mg/m2/day divided BID (days 5 - 33)
  vincristine sulfate: 1.5mg/m2 (max 2 mg) iv push q week (days 5, 12)
Arm/Group | Decitabine / Vorinostat
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine / Vorinostat (N=13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Decreased respiratory rate (Respiratory, thoracic and mediastinal disorders) | 1
Infection, blood (Infections and infestations) | 6
Pain, generalized body (Musculoskeletal and connective tissue disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoxia - acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Lipase elevated (Investigations) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Pain, abdominal (Gastrointestinal disorders) | 1
Hypercholesteremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine / Vorinostat (N=13)
Hemorrhage, bladder (Blood and lymphatic system disorders) | 1
Leukocytes decreased (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 6
Platelets count decreased (Blood and lymphatic system disorders) | 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Bone marrow cellularity (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukocytes (Blood and lymphatic system disorders) | 2
Neutrophils (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 2
Ventricular arrythmia (Cardiac disorders) | 1
Systolic murmur (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Photophobia (Eye disorders) | 1
Blurred vision (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Fluid retention, ascites (Gastrointestinal disorders) | 1
Lower molar pain (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Mucositis (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Edema, lower extremity (General disorders) | 2
Edema, upper extremity (General disorders) | 1
Generalised body aches (General disorders) | 1
Weakness (General disorders) | 1
Fever (General disorders) | 2
Infection, meningitis (Infections and infestations) | 1
Fungal infection, lung (Infections and infestations) | 1
Infection, soft tissue (Infections and infestations) | 1
Infection, neutopenia (Infections and infestations) | 2
Infection, positive blood culture (Infections and infestations) | 1
Pain uncontrolled (Injury, poisoning and procedural complications) | 1
Pain, epigastric (Injury, poisoning and procedural complications) | 1
Pain, headache (Injury, poisoning and procedural complications) | 1
Pain, pedal bilateral (Injury, poisoning and procedural complications) | 1
Pain, leg bilateral (Injury, poisoning and procedural complications) | 2
Pain, stomach (Injury, poisoning and procedural complications) | 1
Pain, left chest (Injury, poisoning and procedural complications) | 1
Pain, low back/leg (Injury, poisoning and procedural complications) | 1
Lower lip swelling (Injury, poisoning and procedural complications) | 1
Pain, NOS (Injury, poisoning and procedural complications) | 1
Hyperbilirubinemia (Investigations) | 4
Weight gain (Investigations) | 1
Creatinine (Investigations) | 1
Lipase elevated (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
ALT increased (Investigations) | 4
Creatinine increased (Investigations) | 2
Fibrinogen increased (Investigations) | 1
Amylase (Investigations) | 1
Lipase (Investigations) | 1
ANC (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Investigations) | 1
AST increased (Investigations) | 1
AST (Investigations) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperchloremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Albumin (Metabolism and nutrition disorders) | 2
Calcium (Metabolism and nutrition disorders) | 2
Glucose (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Uric acid increased (Metabolism and nutrition disorders) | 1
Calcium decreased (Metabolism and nutrition disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 2
Calcium increased (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Somnolence (Nervous system disorders) | 2
Headaches (Nervous system disorders) | 2
Hemiparesis, right side (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 4
Mood alteration, NOS (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infiltrate (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hand foot reaction (Skin and subcutaneous tissue disorders) | 1
Demi Erythema (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Ulceration, decubitus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes